CLINICAL TRIAL: NCT01680380
Title: Tracking Breathing During Sleep With Non-contact Sensors
Status: Withdrawn | Type: Observational
Why Stopped: Superseded by larger funded study
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alexander Kain, Assistant Professor, Oregon Health and Science University
Other Study IDs: IRB00008533
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Sleep Apnea Syndromes; Snoring
Keywords: sleep apnea; snoring
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- At-Home: Overnight sleep at home

SUMMARY:
The purpose of this study is to evaluate the feasibility of tracking breathing during sleep with non-contact sensors (for example, microphones or wireless movement sensors). The investigators will use the data collected with these sensors to develop algorithms for tracking breathing during sleep. The investigators will assess the performance of the algorithms by comparing automatic output against manually-generated labels.

DETAILED DESCRIPTION:
Subjects will be asked to place non-contact sensors (for example, ambient microphones, wireless movement sensors) in their home sleep environment. No sensors will be attached to or otherwise in contact with the subject's body. The subjects will start the data collection before they fall asleep, and stop the data collection the next morning when they wake. The subjects will then return the sensors to the investigator for analysis.

The investigators will study the data and associated manual labeling. The investigators will develop algorithms that use statistical and machine-learning methods to train computer models designed to track breathing automatically. The investigators will compare the automatic output against manually generated labels to determine breath-tracking accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-89
* No self-reported sleep breathing problems

Exclusion Criteria:

* Positive diagnosis for sleep breathing problem (e.g., obstructive sleep apnea)

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the PI's department (OHSU faculty, Ph.D. students) by email and the investigators' personal acquaintances. Participants must be age 21-100 and have no self-reported sleep breathing problems.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Breathing sounds are evident in overnight audio recordings | Night of recording
  This study aims to track breathing during sleep using a high-quality audio interface. Our primary objective is to determine if quiet breathing sounds are visible (in the spectral domain) to trained human labelers.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kain, Ph.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Center for Spoken Language Understanding, Portland, Oregon, United States